CLINICAL TRIAL: NCT06927089
Title: Non-Invasive Hemodynamic Monitoring of Interstitial Lung Disease Patients With Acute Respiratory Failure in Different Modes of Mechanical Ventilation
Brief Title: Non-Invasive Hemodynamic Monitoring of MV ILD Patients With ARF
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Abd El-gayed Eid, Principal Investigator, Assiut University
Other Study IDs: CBBAAS
Record Dates: First submitted 2024-10-25; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Lung Disease (ILD)
Keywords: ILD; MV; non-invasive hemodynamic monitoring
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Non-invasive hemodynamic monitoring of interstitial lung disease (ILD) patients admitted to respiratory ICU with acute respiratory failure and differentiate according to different modes of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Interstitial lung disease patients with acute respiratory failure admitted to respiratory ICU in different modes of MV (NIV, invasive MV and HVNI).

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interstitial lung disease patients with acute respiratory failure admitted to respiratory ICU in different modes of MV (NIV, invasive MV and HVNI).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-16 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Non-invasive Hemodynamic Monitoring | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt